CLINICAL TRIAL: NCT00842075
Title: Effects of Pramlintide in Adolescents With Type 1 Diabetes
Brief Title: Pramlintide in Adolescents With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 05-0724(2)
Record Dates: First submitted 2009-01-20; First posted 2009-02-12 (Estimated); Results first posted 2012-10-19 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2012-09

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; adolescents; post prandial glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — pramlintide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Symlin (Experimental): Subcutaneous injection of pramlintide prior to each meal with reduction of mealtime bolus insulin
  Interventions: Drug: pramlintide
- 2 Usual Regimen (No Intervention): Usual bolus insulin dose at each meal

INTERVENTIONS:
Drug: pramlintide — subcutaneous injection (15 mcg initial dose)prior to meals
  Other Names: Symlin
  Arms: 1 Symlin

SUMMARY:
The investigators hypothesize that subcutaneous pramlintide as an adjunct to mealtime insulin immediately prior to meals can significantly reduce post-prandial glucose concentrations compared with mealtime insulin alone in children with type 1 diabetes.

This is a 36 day, randomized, two-arm, open-label study with a treatment arm (taking pramlintide before all meals) and a control arm (diabetes regimen as usual).

DETAILED DESCRIPTION:
Participants aged 13-17 years who have been diagnosed with type 1 diabetes for more than 1 year will be invited to participate.Other inclusion factors are:

* HbA1c level between 7.5 and 10% inclusive
* Currently using carbohydrate to insulin ratio
* Acceptable form of birth control

Exclusion factors:

* Oral hyperglycemic agents or medications which might affect blood sugar levels
* Recurrent severe hypoglycemia requiring assistance in previous 6 months
* Diagnosis of gastroparesis and/or require use of drugs that stimulate gastrointestinal motility
* Previous use of pramlintide

The study consists of 2 overnight stays at the CTRC where a continuous glucose monitoring system will be worn for twenty-four hours. Blood will be drawn 15 minutes prior to start of each meal and for three hours following each meal. Meals will be controlled for carbohydrate, fat and protein content. Meals will be identical at each CTRC visit.

After a baseline visit for all participants, randomization will occur to either Treatment or Control.Bolus insulin will be adjusted for participants when beginning pramlintide and will likely remain at a reduced rate throughout the trial. All participants will have access to staff to assist with insulin dosing. There will be six mandatory phone visits over the 36 days to ensure the safety of participants in this study.

Insulin, glucose and glucagon levels will be assessed as well as pramlintide levels at final visit of the study. Hypoglycemic events will be tracked, as well as any other adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Between 13 and 17 years of age, inclusive
* Diagnosed with type 1 diabetes for > 1 year
* Hemoglobin A1c between 7.5 and 10% inclusive
* Currently using carbohydrate to insulin ratio
* Acceptable form of birth control

Exclusion Criteria:

* Use of oral hyperglycemic agents or medications affecting blood sugar levels
* Recurrent severe hypoglycemia requiring assistance in past 6 months
* History of hypoglycemia unawareness
* History of gastroparesis requiring use of drugs that stimulate gastrointestinal motility
* Previous use of pramlintide

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2006-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Chase, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Barbara Davis Center, Aurora, Colorado, United States

REFERENCES:
- [Derived] Kishiyama CM, Burdick PL, Cobry EC, Gage VL, Messer LH, McFann K, Chase HP. A pilot trial of pramlintide home usage in adolescents with type 1 diabetes. Pediatrics. 2009 Nov;124(5):1344-7. doi: 10.1542/peds.2008-3750. Epub 2009 Oct 26. PMID 19858155

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 subjects recruited and completed
Pre-assignment Details: no comments
Period: Overall Study
Arm/Group | 1 Symlin | 2 Usual Regimen
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Symlin | 2 Usual Regimen | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 5 | 10
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — study results do not report this | NA (NA) — study results do not report this | 15 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Value After 28 Days
Description: HbA1c values 28 days after randomization
Time Frame: 28
Population: pilot study
Measure: Mean (Standard Deviation); unit: HbA1c %
Arm/Group | 1 Symlin | 2 Usual Regimen
Number analyzed (Participants) | 5 | 5
HbA1c % | 7.94 (0.71) | 8.72 (0.44)

2. Secondary Outcome: Weight Change After 28 Days Intervention Period
Description: Mean weight change after 28 days intervention period
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | 1 Symlin | 2 Usual Regimen
Number analyzed (Participants) | 5 | 5
kg | -0.84 (0.24) | 0.04 (0.62)

ADVERSE EVENTS:
Arm/Group | 1 Symlin | 2 Usual Regimen
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No